CLINICAL TRIAL: NCT03727204
Title: Acute Kidney Injury After Cardiac Surgery: Novel Ultrasound Techniques for Prediction of Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Johan Fridolf Hermansen, Principal Investigator, Aarhus University Hospital
Other Study IDs: 1-10-72-267-18
Record Dates: First submitted 2018-10-09; First posted 2018-11-01 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Acute Kidney Injury; Acute Renal Failure; Cardiac Surgery
Keywords: Ultrasound; Ultrasonographic flow measures; Fluid treatment
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aarhus University Hospital: 100 patients undergoing on-pump cardiac surgery at Charlotte Maxeke Johannesburg Academic Hospital, University of the Witwatersrand
  Interventions: Procedure: On-pump cardiac surgery
- Charlotte Maxeke Johannesburg Academic Hospital, University of the Witwatersrand: 50 patients undergpoing on-pump cardiac surgery at at Charlotte Maxeke Johannesburg Academic Hospital, University of the Witwatersrand
  Interventions: Procedure: On-pump cardiac surgery

INTERVENTIONS:
Procedure: On-pump cardiac surgery — All participants will undergo on-pump cardiac surgery

SUMMARY:
Acute Kidney Injury (AKI) is a frequent and important complication to cardiac surgery. This study will evaluate the diagnostic ability of ultrasonographic measures of blood flow in kidneys and liver in predicting AKI after cardiac surgery.

DETAILED DESCRIPTION:
Acute Kidney Injury (AKI) is a frequent and important complication to cardiac surgery. The pathophysiology is multifactorial, but renal functions in this setting is determined by a complex interplay between renal perfusion, fluid status, cardiac output, mean arterial pressure and back pressure to venous outflow.

Renal perfusion may be quantified with novel ultrasound techniques. Ultrasonography of the kidney and renal vasculature allows for assessment of renal afferent flow and renal venous flow and, together with venous flow patterns of the portal vein and liver veins, may identify patients in risk of AKI.

The study is observational and will describe the diagnostic accuracy of the ultrasound measures in predicting postoperative AKI. Patients will be examined with ultrasound of kidney and liver flow along with echocardiography on on the day before surgery and on the 1st and 4th. In addition, patients are followed with markers of kidney function, fluid balance and invasive measures of mean arterial pressure and central venous pressure.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥ 18 years
* Scheduled for on-pump cardiac surgery
* Oral and written consent

AND

* 1 of the following risk factors for development of postoperative AKI may be included:

  * age > 70 years;
  * NYHA (New York Heart Association) 3+4;
  * Insulin dependent diabetes;
  * Glomerular filtration rate < 60 ml/min/1,73 m2;
  * Ejection fraction < 35;
  * Surgery:

    * Combined CABG and valve surgery;
    * Any valve surgery except isolated aortic-valve surgery;
    * Redo surgery;
    * Endocarditis;
  * Peripheral vascular disease.

Exclusion Criteria:

* Insufficient ultrasonographic imaging of the kidneys;
* Known morphological kidney disease;
* Preoperative dialysis;
* Prior participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for on-pump cardiac surgery at the Department of Cardiothoracic & vascular surgery, Aarhus University Hospital. The study will include 100 patients from Denmark.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
The association between the kidney venous ultrasonography flow pattern category on the 1st postoperative day and acute kidney injury (AKI) on the 4th postoperative day. | 4 days
  The flow pattern is grouped as either continuous, biphasic or monophasic based on the appearance.The final analysis will possibly include other flow categories.
  AKI is defined by the 2012 Kidney Disease: Improving Global Outcomes (KDIGO) criteria and graded in four stages from no AKI to stage 1-3 AKI based on serum creatinin change and/or changes in urine output, with stage 3 being the worst stage.

SECONDARY OUTCOMES:
Correlation between changes in organ-specific flow measurements and the corresponding biomarkers. | 1 month
  Correlations between organ-specific ultrasonography flow measurements and the corresponding biomarkers of kidneys, liver and heart function, for both absolute values of organ-specific flow and perioperative changes in organ-specific flow
Establishment of the most optimal organ specific cut-off values and the development of AKI. | 1 month
  Establishment of the most optimal cut-off (threshold) values for
  * absolute ultrasonography flow values for respectively kidney arterial flow; kidney venous flow; liver vein flow; portal vein flow and the risk of development of AKI.
  * changes in ultrasonography flow values for respectively kidney arterial flow; kidney venous flow; liver vein flow; portal vein flow and the risk of development of AKI.
Fluid balance and AKI | 1 month
  Correlations between accumulated fluid balance on the 1st postoperative day and the development of AKI on the 4th postoperative day.
Diastolic dysfunction and AKI | 1 month
  Correlations between echocardiographic measures of diastolic dysfunction and AKI. The measures include mitral inflow (E and A), mitral annular motion, medial and lateral (e' and a'), and measures define grades of diastolic dysfunction from normal to grade I-III, with grade III being the worst.
Organ-specific flow measures and mortality | 1 month
  Correlation between organ-specific ultrasonography flow measurements on the day before surgery, the 1st and 4th postoperative day and the mortality at the 1st, 4th and 28th postoperative day.
Organ-specific flow measures and and time of stay in ICU and hospital | 1 month
  Correlation between organ-specific ultrasonography flow measurements on the day before surgery, the 1st and 4th postoperative day and the duration of intensive care stay and duration of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Juhl-Olsen, MD, PhD, Study Chair — Department of Anaesthesiology, Aarhus University Hospital
Locations (2):
- Aarhus University Hospital, Department of Anaesthesiology, Aarhus, Denmark
- Department of Anesthesiology, Charlotte Maxeke Johannesburg Academic Hospital, University of the Witwatersrand, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No